CLINICAL TRIAL: NCT07203352
Title: Efficacy and Safety of Targeted Drugs Combined With Chemotherapy in the Treatment of Patients With Newly Diagnosed Acute T-lymphocytic Leukemia
Brief Title: Efficacy of Targeted Drugs Combined With Chemotherapy in the Treatment of T-ALL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2025-241
Record Dates: First submitted 2025-09-23; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): The subjects randomly assigned to the experimental group received targeted drug treatment in addition to the chemotherapy regimen during the second course. Based on the results of bone marrow PCR, subjects with molecular typing of ABL1/ABL2/PDGFRB fusion were to receive chemotherapy combined with dasatinib 100mg orally once a day; subjects with molecular typing of FLT3-ITD positive were to receive chemotherapy combined with sorafenib 400mg orally twice a day.
  Interventions: Drug: targeted drug
- control group (No Intervention): Patients randomly assigned to the control group will receive standard chemotherapy treatment, but they cannot use targeted drugs in combination.

INTERVENTIONS:
Drug: targeted drug — Patients randomly assigned to the control group will receive standard chemotherapy treatment, but they cannot use targeted drugs in combination.The subjects randomly assigned to the experimental group received targeted drug treatment in addition to the chemotherapy regimen during the second course. Based on the results of bone marrow PCR, subjects with molecular typing of ABL1/ABL2/PDGFRB fusion were to receive chemotherapy combined with dasatinib 100mg orally once a day; subjects with molecular typing of FLT3-ITD positive were to receive chemotherapy combined with sorafenib 400mg orally twice a day.
  Arms: experimental group

SUMMARY:
This prospective, randomized, controlled trial evaluates the efficacy and safety of a new targeted drug combined with chemotherapy versus standard chemotherapy alone. Eligible patients were randomized 1:1 to either the treatment or control group.

DETAILED DESCRIPTION:
This study is a prospective, randomized, controlled clinical trial aimed at evaluating the efficacy and safety of the new targeted drug combined with chemotherapy. After signing the informed consent form, patients who met the inclusion/exclusion criteria were randomly assigned to the treatment group and the control group at a ratio of 1:1. Both groups of subjects received standard induction chemotherapy in the first course. Patients in the treatment group would receive corresponding targeted drug combined chemotherapy based on bone marrow PCR testing, while patients in the control group would receive standard chemotherapy. Both the treatment group and the control group would select subsequent treatments based on the chemotherapy efficacy of the subjects. Each subject would undergo regular bone marrow examinations and other evaluations for the underlying disease on a regular basis.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects were diagnosed with acute T-lymphocytic leukemia (according to the 2016 WHO classification) based on their bone marrow pathology and hematology, and sufficient bone marrow samples were available for PCR analysis;
2. The subjects must have never received anti-leukemia treatment before;
3. Age ≥ 18 years old, gender not restricted;
4. The subjects' Eastern Cooperative Oncology Group (ECOG) performance status score is 0-2;
5. The subjects or their legal representatives must provide written informed consent before undergoing the special examinations or procedures of the study.

Exclusion Criteria:

1. Classified as other types of leukemia according to the WHO 2016 classification;
2. Previously received systemic or local treatments including chemotherapy;
3. Previously underwent hematopoietic stem cell transplantation;
4. Had other tumors in addition to leukemia;
5. Had uncontrolled cardiovascular and cerebrovascular diseases, coagulation disorders, severe infectious diseases, etc.;
6. Patients with a history of allergic reactions to any drugs in this research protocol;
7. Left ventricular ejection fraction ≤ 50%;
8. Laboratory test values at screening (unless caused by leukemia): ALT or AST higher than twice the upper limit of normal, AKP and bilirubin higher than 1.5 times the upper limit of normal, creatinine level higher than 1.5 times the upper limit of normal;
9. Other concurrent and uncontrolled medical conditions that the researcher considers will affect the patient's participation in the study;
10. Psychiatric patients or other patients known or suspected to be unable to fully comply with the study protocol;
11. Pregnant or lactating women;
12. HIV-infected individuals.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2-year

SECONDARY OUTCOMES:
Progress-free survival | 2-year
Cumulative incidence of relapse | 2-year

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China